CLINICAL TRIAL: NCT06693271
Title: A Randomized Controlled Trial Investigating the Synergistic Effects of Protein, Blueberries, and Exercise on Cardiovascular Health and Frailty in Older Nova Scotians
Brief Title: Investigating the Combined Effects of Protein, Blueberries, and Exercise on Cardiovascular Health and Frailty in Older Nova Scotians
Acronym: STRONG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University, Canada (Unknown)
Responsible Party: Principal Investigator, Scott Grandy, Associate Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STRONG_2024-2027
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Disease; Frailty
Keywords: Cardiovascular Disease; Frailty; Blueberries; Exercise; Protein; Obesity; Hypertension; Hyperlipidemia; Sedentary Lifestyle; Older Adults
MeSH Terms: conditions — Cardiovascular Diseases; Frailty; Motor Activity; Obesity; Hypertension; Hyperlipidemias; Sedentary Behavior | interventions — blueberry extract; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention of protein, blueberries, and exercise (Active Comparator): treatment groups will receive the STRONG intervention of 30g/day (1 scoop) of a colorless, tasteless whey protein isolate powder supplement and 1 cup (150 grams) of blueberries per day. They will also participate in three 60-minute multimodal exercise sessions per week. Each session will include a warm-up and cool-down (~5 minutes each), 30 minutes of moderate intensity aerobic exercise and 20 minutes of moderate intensity resistance training.
  The intervention lasts for 12 months.
  Interventions: Dietary Supplement: intervention of protein, blueberries; Behavioral: Exercise training
- Control group (No Intervention): Participants receive usual standard of care.

INTERVENTIONS:
Dietary Supplement: intervention of protein, blueberries — intervention of 30g/day (1 scoop) of a colorless, tasteless whey protein isolate powder supplement and 1 cup (150 grams) of blueberries per day.
  Arms: intervention of protein, blueberries, and exercise
Behavioral: Exercise training — Three 60-minute multimodal exercise sessions per week. Exercise interventions will be individualized to each participant based on their fitness level as per recommended guidelines for older adults. Each session will include a warm-up and cool-down (~5 minutes each), 30 minutes of moderate intensity aerobic exercise and 20 minutes of moderate intensity resistance training.
  Arms: intervention of protein, blueberries, and exercise

SUMMARY:
Cardiovascular diseases (CVD) are a leading cause of morbidity and mortality worldwide. While CVDs are predominantly diseases of aging, age itself does not predict CVD risk; people age at different rates. Frailty is a state of accelerated aging that increases the risk of adverse health outcomes. Frail people are at higher risk of developing CVDs, experiencing complications, and dying from these diseases than fit people of the same age. Indeed, frailty predicts the likelihood of developing CVD independently of traditional risk factors for CVD. It is known that older women are frailer than men and tend to express CVDs differently than men, but whether relationships between frailty and CVD are sex specific is unclear. It is possible that shared pathophysiological mechanisms such as chronic inflammation may help explain links between CVD and frailty. Importantly, the degree of frailty can be modified by lifestyle interventions. For example, sedentary lifestyles, food insecurity, and suboptimal dietary habits can exacerbate frailty whereas diet and exercise interventions can attenuate frailty.

The investigators propose that a comprehensive health strategy targeting diet and physical activity to reduce frailty will reduce the risk of cardiovascular disease (CVD), thereby promoting healthy aging. Engaging in physical activity (e.g. exercise) helps improve aerobic fitness, increase muscle mass, promote cardiac regeneration, enhance metabolic function, regulate blood pressure, improve insulin sensitivity, reduce inflammation (a key frailty mechanism), and lessen frailty. High-quality dietary protein is essential to maintain muscle mass/function, preserve mobility, attenuate inflammation, and reduce frailty. Packed with antioxidants such as anthocyanins and flavonoids, with high levels of fiber, vitamins, and minerals, blueberries, a local Nova Scotian food, can help lower blood pressure, improve blood vessel function, reduce inflammation, and help the body utilize dietary protein. These are critical aspects of a strong heart and healthy aging. To date, many frailty intervention studies have been limited by small sample sizes, underrepresentation of women, and/or by testing individual lifestyle modifications rather than synergistic effects; additionally, none have investigated how reducing frailty impacts cardiovascular outcomes. Our goal is to determine if a year-long multidomain intervention of protein, blueberries, and exercise reduces frailty and cardiovascular disease risk in older at-risk Nova Scotians of both sexes.

DETAILED DESCRIPTION:
The proposed trial is a randomized control trial (RCT) investigating the synergistic effects of protein, blueberries, and resistance plus aerobic training on frailty and cardiovascular health in at-risk Nova Scotians. As frailty and CVD are closely linked, the investigators propose that lifestyle interventions to reduce frailty will improve cardiovascular health in at risk individuals. Studies designed to reduce frailty to date are limited by testing individual lifestyle modifications rather than a prescribed package combining theoretically synergistic treatments and none have investigated effects on cardiovascular health. The investigators have developed a novel packaged intervention of exercise plus protein and blueberries based on their effectiveness as individual treatments and potential for synergy based on complementary biological mechanisms. The investigators will determine whether this prescribed STRONG intervention reduces frailty and improves cardiovascular health in older Nova Scotians by comparing the treatment group with a control group who will receive their usual medical care, as in most pragmatic trials that are performed to determine if an intervention can improve current practice. Usual medical care may differ between participants; it may or may not include diet and exercise recommendations from their physicians. The trial design for the STRONG study is a pragmatic randomized controlled trial on year in length with an additional year of follow-up. The participants will be randomly assigned to one of two groups for 12 months: the control group (n=120 who will receive usual care), or the treatment group (n=120; who will receive the STRONG intervention of protein, blueberries, and exercise). The control group will be tested for fitness, frailty, and cardiovascular health including blood biomarkers and cardiac function (echocardiography). They will be given 'report cards' with their test results to monitor their health; the treatment group will receive the reports cards as well. Exercise intensity will be monitored using the Category Ratio 10 (CR10) ratings of perceived exertion scale. On this scale, exercise should elicit a score of 4-5. All participants will be given a copy of the CR10 scale and taught how to use it. The exercise prescription will be individualized to each participant based on their pre-intervention fitness level, level of frailty and medical history. Progression of the program will be determined on an individual basis. All exercise programs will be designed and supervised by a clinical exercise physiologist. A hybrid approach will be used for the exercise sessions. The participant must attend the first exercise session in person and then can choose to attend subsequent sessions in person (Exercise Lab, Dickson Bldg) and/or virtually. All virtual sessions will be delivered via a secure Nova Scotia Health Zoom link. Having the first session in person gives all participants the opportunity to learn and discuss the exercises in a one-on-one format with the clinical exercise physiologist. After the first session it is expected that there may be multiple study participants in in-person or virtual exercise sessions. It is hypothesized that the addition of blueberries to a regimen of exercise plus protein will have synergistic beneficial effects on frailty and cardiovascular health in older individuals.

Our objectives are:

1. To determine whether the STRONG intervention reduces frailty equally in both sexes.
2. To determine whether this intervention improves cardiovascular health in males and females.
3. To determine whether beneficial effects of this intervention are mediated, in part, by effects on markers of chronic inflammation and whether these effects are sex specific

ELIGIBILITY:
Inclusion Criteria:

* Must be between 65 and 85 years of age
* Have at least one cardiovascular risk factor
* Must be able to participate moderate intensity exercise program

Exclusion Criteria:

* Medical and cognitive conditions that prevent participation in the intervention
* Allergies and or dislike of blueberries and/or protein powder

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Fitness | Baseline, 3,6,9, and 12 months
  Assessed using a 6-minute walk test (6MWT). Total distance in meters will be recorded.
Echocardiography | Baseline, 12 Months
  Ejection fraction will be measured in M-mode and global longitudinal strain will be assessed.
Inflammatory Markers | Baseline, 12 Months
  Plasma will be obtained from blood samples collected at two time points, pre- and post-intervention. A multiplex assay will be used to quantify anti-inflammatory and inflammatory cytokines in the plasma sample. The following cytokines will be quantified (pg/ml): APRIL / TNFSF13, BAFF / TNFSF13B, sCD30 / TNFRSF8, sCD163, Chitinase-3-like, gp130 / sIL-6Rβ, IFN-α2, IFN-β, IFN-γ, IL-2, sIL-6Rα, IL-8, IL-10, IL-1, IL-12 (p40), IL-12 (p70), IL-19, IL-20, IL-22, IL-26, IL-27 (p28), IL-28A / IFN-λ2, IL-29/IFN-λ1, IL-32, IL-34, IL-35, LIGHT / TNFSF14, MMP-1, MMP-2, MMP-3, Osteocalcin, Osteopontin, Pentraxin-3, sTNF-R1, sTNF-R2, TSLP, TWEAK / TNFSF12.
Frailty | Baseline, 3,6,9, and 12 months
  Frailty will be assessed using the Clinical Frailty Scale (CFS), Pictorial Fir-Frail Scale (PFFS), and Frailty Index
Cardiovascualr Risk: Blood pressure | Baseline, 3, 6, 9, 12 months
  Resting blood pressure (systolic/diastolic) will be assessed using an automated blood pressure cuff. Blood pressure will be measure in mm of Hg.
Cardiovascualr Risk: Lipid Profile | Baseline, 12 months
  Blood will be drawn by venipuncture and then sent to the hospital lab. There the lipid profile will be determined. Specifically, total cholesterol (mmol/L), triglycerides (mmol/L), low density lipoprotein (mmol/L) and high density lipoprotein (mmol/L) will be quantified.
Cardiovascualr Risk: Blood glucose | Baseline, 12 months
  After fasting for 12 hours the participants blood will be drawn by venipuncture. Blood samples will be sent to the hospital lab and fasting glucose (mmol/L) will be assessed.
Frailty: Clinical Frailty Scale (CFS) | Baseline, 3, 6, 9, 12 months
  Frailty will be assessed using the CFS. The scale for the assessment ranges from 0 to 9, where 0 represents a robust individual and 9 represents terminally ill. A score of 4 or higher indicates frailty. This is a clinical judgement tool.
Frailty: Pictorial Fit to frail Scale (PFFS) | Baseline, 3, 6, 9, 12 months
  Frailty will be assessed with the PFFS. The PFFS is completed by the participant and uses visual images to assess their level of fitness/frailty. There are 14 sets of images on the PFFS. Each set contains 3-4 images and the participant is asked to pick the images that represents how they "usually" feel. The questionnaire is scored out of 43, with higher scores representing a higher degree of frailty.

SECONDARY OUTCOMES:
Muscular Health: Lower Body Strength | Baseline, 3,6,9, and 12 months
  Lower body strength will be assessed using the 30 second sit to stand task. The number of times an individual can stand from a seated position will be recorded.
Balance | Baseline, 3,6,9, and 12 months
  Single leg balance test. Total time in seconds will be recorded.
Mobility: Lower Body | Baseline, 3,6,9, and 12 months
  Lower body mobility will be assessed using the sit & reach test. Reach distance will be measured in centimeters.
Overall Health | Baseline, 3,6,9, and 12 months
  Overall health status will be assessed using the Short-Form 36 Health Survey (SF-36) . The SF-36 contains 10 items. The scores range from 0 to 100, with lower scores representing more disability and higher scores representing less disability.
Muscular Health: Upper Body | Baseline, 3, 6, 9, 12 months
  Upper body strength will be assessed using a hand grip dynamometer. Grip strength will be measured in kg.
Mobility: Upper Body | Baseline, 3, 6, 9, and 12 months.
  Upper body mobility using the shoulder girdle mobility test. The range of motion will be measured in centimeters.

OTHER OUTCOMES:
Safety Outcomes | Safety will be assessed at 1,3,6,9, and 12 months.
  Safety outcomes will be determined by recording the total number of adverse events that occur over the duration of the exercise program. This will be divided by the number of participant hours to determine the number of adverse events/participant hours.
Study Adherence | On the last day of the month particpants will upload the months logbook. (e.g. On November 30th, participant would upload the November logbook). This will be done for every month the participant is in the study (i.e. 12 months).
  Exercise attendance and blueberry/protein consumption will be monitored using an electronic participant logbook.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dickson Building, Halifax, Nova Scotia
  - QEII Health Sciences Centre, Dickson Building, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No